CLINICAL TRIAL: NCT00212498
Title: Tuberculosis Research Blood Bank
Status: Withdrawn | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11354 (previously 4424)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- TB diagnosis
  Interventions: Procedure: Develop a bank of blood samples from patients infected with TB for future molecular genetics studies and serological studies

INTERVENTIONS:
Procedure: Develop a bank of blood samples from patients infected with TB for future molecular genetics studies and serological studies — Blood sample

SUMMARY:
To create a Tuberculosis Research Blood Bank for future molecular genetics and serological studies

ELIGIBILITY:
Inclusion Criteria:

* TB suspect with positive sputum smear

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TB patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Develop TB Blood Bank | Long-Term
  To develop a bank of blood samples (serum, plasma, buffy coat DNA) and urine from patients infected with TB. This blood and urine will be used for future molecular genetics studies. Demographic data will be collected and samples will be stored by number. The banked specimens will be evaluated in an attempt to identify susceptibility genes in TB disease. Specifically, expression of the human Bcg gene that codes for resistance to M. tuberculosis will be evaluated and its expression correlated expression with gender, race, clinical TB characteristics. Each patient will have a unique identifier and therefore data generated from this analysis will not be linkable to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rany Condos, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine Division of Pulmonary and Critical Care Medicine, New York, New York, United States